CLINICAL TRIAL: NCT00365872
Title: Combination of External Beam Radiation With Intratumoral Injection of Dendritic Cells as Neo-adjuvant Treatment of High-risk Soft Tissue Sarcoma Patients
Brief Title: External Beam Radiation With Intratumoral Injection of Dendritic Cells As Neo-Adjuvant Treatment for Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Cancer Treatment Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14497
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2013-06

CONDITIONS: Soft Tissue Sarcoma
Keywords: Sarcoma; Intratumoral injection; Dendritic cells; Neo-adjuvant treatment; Immunotherapy; Pheresis; Radiation
MeSH Terms: conditions — Sarcoma | interventions — Injections; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBRT + DC Injection + Resection (Experimental): Single Arm: EBRT + DC Injection + Resection. Prior to the fourth DC Injection, participants were assigned to 3 cohorts as outlined in that intervention.
  Interventions: Biological: Dendritic Cell (DC) Injections; Procedure: Radiation therapy; Procedure: Complete Resection - Surgery for tumor removal

INTERVENTIONS:
Biological: Dendritic Cell (DC) Injections — * DCs (10^7 cells) were injected intratumorally three times on the second, third, and fourth Friday during the course of radiation.
  * One additional DC injection was given before surgery to assess DC migration
  * Patients were assigned to one of three cohorts:
  Group 1 - DC injection # 4 given 24 hours prior to surgery Group 2 - DC injection # 4 given 48 hours prior to surgery Group 3 - DC injection # 4 given 72 hours prior to surgery
Procedure: Radiation therapy — Radiation was delivered 5 days per week (Monday-Friday).
Procedure: Complete Resection - Surgery for tumor removal — Tumors were surgically resected 3-6 weeks after the completion of EBRT.

SUMMARY:
This is a Phase II study using a combination of external beam radiation with intratumoral injection of dendritic cells (white blood cells) as neo-adjuvant treatment for patients with high-risk soft tissue sarcoma. The purpose was to determine if an injection of the patient's own immune related white blood cells into their tumor would strengthen the immune system to fight against their cancer.

DETAILED DESCRIPTION:
Patients were treated with external beam radiation therapy (EBRT) combined with experimental intratumoral injection of dendritic cell (DC). Patients received 5,040 centigray (cGy) EBRT in 28 equal fractions. Radiation was delivered 5 days per week (Monday-Friday). DCs (10^7 cells) were injected intratumorally three times on the second, third, and fourth Friday during the course of radiation. One additional DC injection was given several days before surgery to assess DC migration. Tumors were surgically resected 3-6 weeks after the completion of EBRT.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate or high grade sarcoma as determined by pathology review
* Musculoskeletal tumor in extremities, trunk or chest wall.
* Primary tumor or isolated locally recurrent tumor greater than 5 cm in diameter.
* Clinical Stage T2N0M0 (AJCC 6th edition)
* Patient is not a candidate for neoadjuvant chemotherapy.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* No steroid therapy within 4 weeks of first dendritic cell administration.
* No coagulation disorder.
* Patient's written informed consent.
* No contraindication to resection.
* Adequate organ function (measured within a week of beginning treatment).

  * White blood count (WBC) > 3,000/mm to the third power and absolute neutrophil count (ANC) >1500/mm to the third power
  * Platelets > 100,000/mm to the third power
  * Hematocrit > 25%
  * Bilirubin < 2.0 mg/dL
  * Creatinine < 2.0 mg/dL, or creatinine clearance > 60 mL/min
* Radiation Oncologist must confirm that a 2-3 cm strip of skin can be spared from radiation.

Exclusion Criteria:

* Retroperitoneal location.
* Gastrointestinal stromal tumor (GIST).
* Demonstrated metastatic disease.
* Prior radiation therapy if the current tumor is locally recurrent after prior resection.
* Concurrent treatment with any anticancer agent other than radiation as dictated by the protocol.
* Bleeding disorder.
* H.I.V. infection or other primary immunodeficiency disorder.
* Ongoing systemic therapy with immunosuppressant drugs (e.g. corticosteroids, azathioprine, cyclosporin, methotrexate).
* Any serious ongoing infection.
* Pregnant or lactating women -- Patients in reproductive age must agree to use contraceptive methods for the duration of the study (a pregnancy test will be obtained before treatment).
* ECOG performance status of 2, 3 or 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Antonia, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Hong WX, Sagiv-Barfi I, Czerwinski DK, Sallets A, Levy R. Neoadjuvant Intratumoral Immunotherapy with TLR9 Activation and Anti-OX40 Antibody Eradicates Metastatic Cancer. Cancer Res. 2022 Apr 1;82(7):1396-1408. doi: 10.1158/0008-5472.CAN-21-1382. PMID 35135810
- [Derived] Raj S, Bui MM, Springett G, Conley A, Lavilla-Alonso S, Zhao X, Chen D, Haysek R, Gonzalez R, Letson GD, Finkelstein SE, Chiappori AA, Gabrilovitch DI, Antonia SJ. Long-Term Clinical Responses of Neoadjuvant Dendritic Cell Infusions and Radiation in Soft Tissue Sarcoma. Sarcoma. 2015;2015:614736. doi: 10.1155/2015/614736. Epub 2015 Dec 31. PMID 26880867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with histologically confirmed large high grade soft-tissue sarcomas (STS) of the extremity/trunk/chest wall were enrolled to the study from 5/18/2006 to 2/19/2009. These patients had clinical stage T2N0M0 with a significant (>50%) risk of progressing to distant metastases.
Groups:
- COHORT 1: EBRT + DC Injection + Resection; COHORT 2: EBRT + DC Injection + Resection; COHORT 3: EBRT + DC Injection + Resection: Single Arm: EBRT + DC Injection + Resection. Prior to the fourth DC Injection, participants were assigned to 3 cohorts for that injection only.
  Dendritic Cell (DC) Injections: DCs (10^7 cells) were injected intratumorally three times on the second, third, and fourth Friday during the course of radiation. One additional DC injection was given before surgery to assess DC migration. Patients were assigned to one of three cohorts: Group 1 - DC injection # 4 given 24 hours prior to surgery, Group 2 - DC injection # 4 given 48 hours prior to surgery, Group 3 - DC injection # 4 given 72 hours prior to surgery.
  Radiation was delivered 5 days per week (Monday-Friday). Complete Resection - Surgery for tumor removal: Tumors were surgically resected 3-6 weeks after the completion of EBRT.
Period: Overall Study
Arm/Group | COHORT 1: EBRT + DC Injection + Resection | COHORT 2: EBRT + DC Injection + Resection | COHORT 3: EBRT + DC Injection + Resection
Started | 5 | 6 | 6
Completed | 5 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All evaluable participants available for follow-up at time of analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | COHORT 1: EBRT + DC Injection + Resection | COHORT 2: EBRT + DC Injection + Resection | COHORT 3: EBRT + DC Injection + Resection | Total
Number analyzed (Participants) | 5 | 6 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 3 | 11
  >=65 years | 0 | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 35 [25 to 53] | 61 [41 to 81] | 68 [55 to 81] | 53 [25 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 4 | 5 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Immune responses in patients treated with EBRT and DCs: Transient immune response = response detected at only one time point; Robust immune response = response detected at least at two time points. An individual patient was considered a responder to tumor cell lysates (TCL) or survivin if at any time point the response in the interferon gamma (IFN-γ) enzyme-linked immunospot (ELISPOT) assay was higher than 30 spots per 2 X 10^5 cells and in the proliferation assay higher than 3,000 counts per minute (CPM) and the response in IFN-γ ELISPOT or proliferation assays to TCL or Ad-surv was more than 2 standard deviations (SD) higher than the response to the corresponding control lysate or Ad-c at the same time point and 2 SD higher than the response to the same stimuli before start of the treatment.
Time Frame: Up to 3 years
Population: All evaluable participants available for follow-up at time of analysis.
Measure: Number; unit: participants
Groups:
- EBRT + DC Injection + Resection: Single Arm: EBRT + DC Injection + Resection. Prior to the fourth DC Injection, participants were assigned to 3 cohorts for that injection only.
  Dendritic Cell (DC) Injections: DCs (10^7 cells) were injected intratumorally three times on the second, third, and fourth Friday during the course of radiation. One additional DC injection was given before surgery to assess DC migration. Patients were assigned to one of three cohorts: Group 1 - DC injection # 4 given 24 hours prior to surgery, Group 2 - DC injection # 4 given 48 hours prior to surgery, Group 3 - DC injection # 4 given 72 hours prior to surgery.
  Radiation was delivered 5 days per week (Monday-Friday).
  Complete Resection - Surgery for tumor removal: Tumors were surgically resected 3-6 weeks after the completion of EBRT.
Arm/Group | EBRT + DC Injection + Resection
Number analyzed (Participants) | 17
participants
  Developed Tumor Specific Response | 9
  Transient Response | 3
  Robust Response | 6

2. Secondary Outcome: Occurrence of Significant (>/= Grade 2) Toxicity
Description: Toxicity assessment during combination external beam radiation therapy (EBRT)/DC neoadjuvant treatment. Toxicity was assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 criteria.
Time Frame: Up to 3 years
Population: All evaluable participants available for follow-up at time of analysis.
Measure: Number; unit: participants
Arm/Group | EBRT + DC Injection + Resection
Number analyzed (Participants) | 17
participants | 0

3. Secondary Outcome: Occurrence of Postoperative Wound Complications
Description: Postoperative wound complications were defined using NCI Common Toxicity Criteria (CTC).
Time Frame: Up to 3 years
Population: All evaluable participants available for follow-up at time of analysis.
Measure: Number; unit: participants
Arm/Group | EBRT + DC Injection + Resection
Number analyzed (Participants) | 17
participants | 5

4. Secondary Outcome: Participants With No Evidence of Disease at Follow-up
Description: Participants who had no evidence of the disease for at least one year after the start of the treatment (time of follow-up); for at least 2 years, and for at least 3 years.
Time Frame: 3 years
Population: All evaluable participants available for follow-up at time of analysis.
Measure: Number; unit: participants
Arm/Group | EBRT + DC Injection + Resection
Number analyzed (Participants) | 17
participants
  At One Year Follow-up | 12
  At Two Year Follow-up | 6
  At Three Year Follow-up | 4

5. Other Pre Specified Outcome: Number of Participants With Increase in Level of Radioactivity at Excision Per Cohort
Description: To identify the nodes to be excised, an injection with Indium 111 (radio active dye) labeled dendritic cells (of vaccine #4) was performed 1 to 3 days prior to surgery. Patients were evenly divided to be assigned to one of three cohorts: Cohort 1, 1 day before surgery; Cohort 2, 2 days before surgery; Cohort 3, 3 days before surgery. Vaccine #4 was labeled in order to evaluate how long dendritic cells need to travel to regional draining lymphatics. Tumor resection was not delayed by this.
Time Frame: Up to 3 years
Population: Participants evaluable for this measure
Measure: Number; unit: participants
Groups:
- Single Arm - Cohort 1: DC injection # 4 given 24 hours prior to surgery
- Single Arm - Cohort 2: DC injection # 4 given 48 hours prior to surgery
- Single Arm - Cohort 3: DC injection # 4 given 72 hours prior to surgery
Arm/Group | Single Arm - Cohort 1 | Single Arm - Cohort 2 | Single Arm - Cohort 3
Number analyzed (Participants) | 5 | 4 | 6
participants | 0 | 4 | 6

ADVERSE EVENTS:
Time Frame: 3 years
Description: All participants
Arm/Group | EBRT + DC Injection + Resection
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBRT + DC Injection + Resection (N=17)
Wound complication, non-infectious - Possibly related (Skin and subcutaneous tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue, Other - Unrelated (Musculoskeletal and connective tissue disorders) | 1 (1)
Dermatology/Skin, Other - Unrelated (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral arterial ischemia - Unrelated (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism - Unrelated (Vascular disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, Wound - Probably related (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EBRT + DC Injection + Resection (N=17)
Fatitue (General disorders) | 1
Constitutional Symptoms - Other (General disorders) | 4
Insomnia (General disorders) | 3
Rigors/chills (General disorders) | 2
Weight loss (Metabolism and nutrition disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 1
Pain - Other (General disorders) | 11
Pain - Extremity-limb (General disorders) | 8
Pain - Head/headache (General disorders) | 4
Pain - Back (General disorders) | 3
Pain - Joint (General disorders) | 3
Pain - Abdomen NOS (General disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 1
Pain - Stomach (General disorders) | 1
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 3
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 3
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 2
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 10
Anorexia (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Mood alteration - Anxiety (General disorders) | 3
Neurology - Other (General disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 2
Dizziness (General disorders) | 1
Mood alteration - Depression (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-upper (Musculoskeletal and connective tissue disorders) | 1
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1
Edema: limb (Blood and lymphatic system disorders) | 4
Lymphatics - Other (Blood and lymphatic system disorders) | 1
Vision-Blurred vision (Eye disorders) | 2
Ocular/Visual - Other (Eye disorders) | 1
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Allergy/Immunology - other (Immune system disorders) | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1
Infection with unknown ANC - Wound (Infections and infestations) | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Hypertension (Cardiac disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 1
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes